CLINICAL TRIAL: NCT01959009
Title: Does High Frequency Oscillatory Ventilation Combined With Intermittent Sigh Breaths Improve Oxygenation Compared to High Frequency Oscillatory Ventilation Without Sigh Breaths in Neonates?
Brief Title: High Frequency Oscillatory Ventilation Combined With Intermittent Sigh Breaths: Effects on Blood Oxygenation and Stability of Oxygenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christian Heiring, Neonatologist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-2-2012-167
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Respiratory Distress Syndrome, Newborn; Bronchopulmonary Dysplasia; Ventilator Induced Lung Injury
Keywords: newborn, lung disease, mechanical ventilation, lung recruitment, high frequency ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Bronchopulmonary Dysplasia; Ventilator-Induced Lung Injury; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFOV-sigh at start (Experimental): Each patient will be exposed to either HFOV alone (HFOV-only) or HFOV combined with sigh breaths (HFOV-sigh), but in different order.
  MAP=mean airway pressure.
  DURING HFOV-SIGH:
  * Frequency 3 breaths/min
  * Ti = 1s
  * Peak inspiratory pressure (PIP) = 30 cm H2O
  For patients already on HFOV-sigh at study start:
  • MAP-set will be left unchanged at pre-trial settings.
  For patients on HFOV-only at study start:
  • During periods with superimposed sigh breaths, MAP-set will be reduced in accordance with a calculation of MAP aiming to keep average mean airway-pressure (MAP) unchanged. (MAP=(PIP*Tinsp+PEEP*Texp)/(Tinsp+Texp)
  DURING HFOV-ONLY
  For patients on HFOV-sigh at study start:
  • During HFOV-only, the MAP-set will be increased in accordance with a calculation of MAP, aiming to keep average mean airway-pressure (MAP) unchanged.
  For patients on HFOV-only at study start:
  • MAP-set will be left unchanged at pre-trial settings.
  Interventions: Other: HFOV combined with sigh breaths
- HFOV-only at start (Experimental): Each patient will be exposed to either HFOV alone (HFOV-only) or HFOV combined with sigh breaths (HFOV-sigh), but in different order.
  MAP=mean airway pressure.
  DURING HFOV-SIGH:
  * Frequency 3 breaths/min
  * Ti = 1s
  * Peak inspiratory pressure (PIP) = 30 cm H2O
  For patients already on HFOV-sigh at study start:
  • MAP-set will be left unchanged at pre-trial settings.
  For patients on HFOV-only at study start:
  • During periods with superimposed sigh breaths, MAP-set will be reduced in accordance with a calculation of MAP aiming to keep average mean airway-pressure (MAP) unchanged. (MAP=(PIP*Tinsp+PEEP*Texp)/(Tinsp+Texp)
  DURING HFOV-ONLY
  For patients on HFOV-sigh at study start:
  • During HFOV-only, the MAP-set will be increased in accordance with a calculation of MAP, aiming to keep average mean airway-pressure (MAP) unchanged.
  For patients on HFOV-only at study start:
  • MAP-set will be left unchanged at pre-trial settings.
  Interventions: Other: HFOV combined with sigh breaths

INTERVENTIONS:
Other: HFOV combined with sigh breaths — We plan only to investigate infants already ventilated on the HFOV-modus on high frequency oscillators, where the HFOV modus can be superimposed on conventional modes of ventilation. This gives the opportunity to combine HFOV with intermittent sigh breaths with a pre-set frequency and pre-set peak inspiratory pressure (PIP) and thus comparing HFOV combined with sigh breaths (HFOV-sigh) with conventional HFOV (HFOV-only).
  All included participants will be exposed to the two different ventilator strategies tested in this trial, albeit in alternating and different order.
  Each patient will serve, as it's own control. The trial will involve four alternating 1-hours periods allowing a sufficient "wash-out" period, as it has been shown that alveolar recruitment and derecruitment may take up to 25 min after changes to ventilator pressures At study start the patients will randomly be assigned to either starting with HFOV-only or HFOV-sigh

SUMMARY:
Background:

Ventilator induced lung injury (VILI) remains a problem in neonatology. High frequency oscillatory ventilation (HFOV) provides effective gas exchange with minimal pressure fluctuation around a continuous distending pressure and therefore small tidal volume. Animal studies showed that recruitment and maintenance of functional residual capacity (FRC) during HFOV ("open lung concept") could reduce lung injury.

"Open lung HFOV" is achieved by delivering a moderate high mean airway pressure (MAP) using oxygenation as a guide of lung recruitment. Some neonatologists suggest combining HFOV with recurrent sigh-breaths (HFOV-sigh) delivered as modified conventional ventilator-breaths at a rate of 3/min. The clinical observation is that HFOV-sigh leads to more stable oxygenation, quicker weaning and shorter ventilation. This may be related to improved lung recruitment. This has however to our knowledge not been tested in a clinical trial using modern ventilators.

Purpose, aims:

* To compare HFOV-sigh with HFOV-only and determine if there is a difference in oxygenation expressed as a/A-ratio and/or stability of oxygenation expressed as percentage time with oxygen saturation outside the reference range.
* To provide information on feasibility and treatment effect of HFOV-sigh to assist planning larger studies. We hypothesize that oxygenation is better during HFOV-sigh.

Methods:

Infants at 24-36 weeks corrected gestational age already on HFOV are eligible. Patients will be randomly assigned to HFOV-sigh (3 breaths/min) followed by HFOV-only or vice versa for 4 alternating 1-hours periods (2-treatment, double crossover design, each patient being its own control). During HFOV-sigh set-pressure will be reduced to keep MAP constant, otherwise HFOV will remain at pretrial settings. Outcome will be calculated from normal clinical parameters including pulx-oximetry and transcutaneous monitoring of oxygen and carbon-dioxide partial pressures.

DETAILED DESCRIPTION:
High frequency oscillatory ventilation (HFOV) has been used in neonatal respiratory care for more than three decades. HFOV provides effective gas exchange with minimal pressure fluctuation around a set mean airway pressure (MAP) functioning as a continuous distending pressure (CDP), and low tidal volume compared to conventional ventilation (CV). HFOV was therefore thought to be able to reduce the risk of bronchopulmonary dysplasia in ventilated preterm babies. However results from randomized controlled trials comparing HFOV with conventional ventilation have been conflicting and meta-analyses have not shown clear evidence that HFOV is safer or more effective than conventional ventilation neither when used as initial strategy nor as rescue strategy in preterm babies with respiratory distress syndrome (RDS). Consequently there are no absolute indications for HFOV in preterm babies and most neonatologists today use HFOV as a rescue mode when conventional ventilation is failing in the acute setting of RDS as well as in the baby with bronchopulmonary dysplasia.

Maintaining adequate functional residual capacity (FRC) together with the fraction of inspired oxygen FiO2 are the main determinants of oxygenation. The larger the FRC, the larger is the volume of available oxygen in the alveoli for gas transport. Adequate oxygen saturation (SAT) of the blood in room air or an improvement in oxygen-saturation without changing the fraction of inspired oxygen can be seen as an indirect indicator of normal or normalized FRC, and most neonatologists use oxygenation as an indirect marker for lung volume during HFOV.

The CDP or set-MAP is the main determinant of lung-aeration during HFOV. A too low MAP may cause non-homogenous aeration and atelectasis leading to atelectotrauma and redirection of airflow to more compliant alveoli leading to localized hyperinflation.

Accordingly, early animal studies showed that recruitment and maintenance of FRC during HFOV could reduce lung injury. Lung recruitment was initially achieved by superimposing conventional ventilation (CV) breaths on top of HFOV with lower MAP than used today, either as recurrent sustained inflations lasting 15-20 seconds about every 20 minute, as intermittent sigh breaths (3-5 tidal breaths pr minute) delivered as normal conventional breaths or as conventional ventilation at normal rate combined with HFOV.

Today most neonatologists perform this so-called "open lung" concept by adjusting the set-MAP using oxygenation as an indirect guide of lung recruitment. Different approaches are used explained by difficulties in direct bedside monitoring of FRC. Some initiate HFOV with MAP 2-3 cm H2O above the MAP needed during conventional ventilation subsequently adjusting MAP until the fraction of inspired O2 (FiO2) <0.25-0.6 providing no signs of over inflation of the lungs on x-ray. Others go through a more complex step-wise increase in MAP till FiO2 cannot be reduced further, and then gradually decrease MAP until FiO2 again needs to be increased to maintain a predefined SAT and then continues ventilations with a MAP set at 2 cm H2O above this point, thereby placing ventilation on the more compliant deflation limb of the pressure-volume relationship of the lung.

During HFOV, MAP may be adjusted as mentioned above. Further increase in MAP may increase FRC by increased aeration and consequently improve oxygenation. Although recent clinical trials suggest this approach is safe, it could potentially lead to generalized hyperinflation and volutrauma in addition to interfering with systemic venous return and cardiac output especially if not combined with direct monitoring of lung volume which is currently not available in routine clinical care.

Combining intermittent recruitment sigh breaths at a rate of 3-5 breaths/minute with HFOV could be an alternate way of assisting in maintaining or normalizing FRC during which MAP is only increased temporarily and intermittently. This could in theory lead to quicker weaning in MAP, less oxygen exposure and potentially reduced lung injury. A concern however could be, that the intermittent sigh breaths will lead to intermittent excessive pressures in distal airways and to excessive tidal volume and accordingly not be beneficial at all. Nevertheless the approach of combining HFOV and sigh breaths at a low rate seems to be encouraged by a number of neonatologist.

It has however to our knowledge not yet been tested in a controlled human trial.

A search on PubMed revealed no human or animal trials comparing HFOV combined with intermittent recruitment sigh-breaths at a low rate. Also no trials exploring this approach are currently registered on www.clinicaltrials.gov.

To our knowledge so far only one human trial comparing HFVO with recruitment breaths at low rate has been registered but never published (Texas Infant Star Trial).

Combining HFOV with conventional breaths has only been reported in a limited number of studies and only with focus on HFOV combined with CV at normal rate showing a possible benefit. Similar results have been reported when comparing High frequency Jet Ventilation (HFVJ) combined with CV at normal rate with HFVJ alone.

Trial rationale:

Combining intermittent recruitment sigh breaths at a low rate with HFOV could offer a further way of assisting in maintaining or normalizing FRC with only modest or no increase in MAP in alignment with the open lung concept.

A concern however could be, that the intermittent sigh breaths will lead to intermittent increased pressures in distal airways and too large tidal volume and accordingly not be beneficial at all. Despite this, the approach of combining HFOV and sigh breaths seems to be encouraged by a number of neonatologist.

It has however, to our knowledge not yet been tested in a controlled human trial. We therefore wish to conduct a controlled cross-over trial assessing the effect of HFOV combined with intermittent sigh breaths on oxygenation in ventilated neonates using oxygenation as an indirect indicator of lung recruitment.

Objective and hypothesis:

The objectives of this trial are to:

• Compare HFOV combined with intermittent recruitment sigh breaths at a rate of 3/min (HFOV-sigh) with HFOV only (HFOV-only) and examine if:

* oxygenation expressed as a/A-ratio improves with HFOV-sigh

  * a/A-ratio is a measure of oxygenation and calculated as
  * a/A-ratio = paO2/(0,95*FiO2- PaCO2),
  * paO2 and PaCO2 are measured on arterial blood if arterial access is in situ otherwise as transcutaneous values (see further down).
* stability of oxygenation improves with HFOV-sigh

  • expressed as a calculation of the percentage deviation of time spent outside the reference range for oxygen-saturation (SAT) for the given gestational age (AUC - area-under-the-curve) and comparing this with MAP and FiO2.
* Evaluate the possibility of setting up a larger randomized controlled trial We hypothesize that during HFOV-sigh the oxygenation will be improved as well at the stability of oxygenation with less time spent outside the reference range for SAT at an unchanged or lower FiO2

Trial design:

The trial is planned as a 4-period 2-treatment, double crossover clinical trial with each patient being its own control. Patients will be randomly assigned to receive HFOV-Sigh followed by HFOV-only or vice versa for four alternating 1-hours periods.

ELIGIBILITY:
Inclusion Criteria:

* Infants at 24-36 weeks corrected gestational age
* Already ventilated with high frequency ventilation
* Requiring FiO2=21%-70% to maintain adequate oxygen saturation.
* Clinical stable

  o i.e. ventilated on current settings for more than just a few hours with stable but not necessarily normalized blood gases or transcutaneous values and oxygen requirement.
* Parent(s) or guardian able and willing to provide informed consent

Exclusion Criteria:

* Major congenital cardiovascular or respiratory abnormalities.
* The attending neonatologist responsible for the baby considers one of the ventilation modes unsuitable for the infant.
* Poor skin integrity precluding use of transcutaneous monitoring.
* Lack of parental signed written informed consent.
* Parents under 18 years of age.

Ages: 24 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2014-08; Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Delta-a/A-ratio | on study day
  a/A-ratio calculated as a/A-ratio= TcPO2/(0,95*FiO2- TcPCO2) By delta-a/A-ratio means the difference in a/A-ratio between the two modes of ventilation, as an indirect measure of lung recruitment.
stability of oxygen saturation | on study day
  The difference in area-under-the-curve for "out of range" for oxygen saturation (based on accepted general reference ranges for the given gestational age).

SECONDARY OUTCOMES:
FiO2 | on study day
  Difference in fraction of inspired oxygen between the two ventilator modes
Partial pressure of CO2 | on study day
  Difference in transcutaneous pCO2 between the two ventilator modes
heart rate | on study date
  Difference in heart rate between the two ventilator modes
Partial pressure of O2 | on study date
  Difference in partial pressure of oxygen measured transcutaneously between the two ventilator modes

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiring, md, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Neonatology, Rigshospitalet, Copenhagen, Denmark